CLINICAL TRIAL: NCT04562350
Title: XatJove Anoia, as a Tool to Bring Health Services Closer to Teenagers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Principal Investigator, Glòria Saüch Valmaña, PhD, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/137-P
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: mHealth; Telehealth; teenager; health promotion and sexual Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A sample of students aged 12 to 16 years from middle school and high school in the sanitary region of Anoia in the course of 2020-21.
  Interventions: Other: XatJove Anoia Aplication
- Control group (No Intervention): A sample of students aged 12 to 16 years from middle school and high school in the sanitary region of Osona in the course of 2020-21.

INTERVENTIONS:
Other: XatJove Anoia Aplication — All students (age 12-16 years) from middle school and high school in the sanitary region of Anoia, province of Barcelona, will access a Platform ( ABH Health), where the users will enter specific registration data ( age, sex..etc), after every visit the users will be provided with a 6 multiple choice questionary and asked to punctuate in a scale from 1 to 10, the satisfaction of the service provided. Appart from this data, researchers will use a software to register specific Health-related words and classify them as Health-problems. While Osona students will attend face-to-face consultations as usual, apart from this data,Registrations will be reviewed later and specific search techniques and strategies will be coded. A qualitative review will be performed too.
  Arms: Intervention group

SUMMARY:
Programs such as "Salut i Escola" aim to improve the health of teenagers through actions to promote health, prevent risk situations and provide early care for problems related to mental health, emotional health and sexual, drug, alcohol and tobacco use, in collaboration with schools and community health services present in the territory. The massive use of new technologies among adolescents means that health programs have to adapt to this reality. XatJove Anoia offers a secure and completely confidential chat with nursing professionals via mobile without having to download any App. In the age of COVID-19, it is important to reduce the risk of infection caused by contact with health services while minimizing non-essential face-to-face visits.Hypothesis: The use of XatJove can increase teenagers' consultations with nursing professionals at Primary Care Centers.Objectives: To demonstrate that through the use of mobile phones and messaging applications, the number of health consultations in "Salut i Escola" program of the Anoia region increases.Methodology: The study uses a mixed methodology comparing the total number of visits (face-to-face and with XatJove) of the "Salut i Escola" program in the Anoia region during the 2020-2021 academic year with the number of face-to-face visits of the same program in the Osona region.Determinations: Number of total consultations in the "Salut i Escola" program during the 2020-2021 academic year in Anoia and Osona. XatJove user satisfaction survey.

DETAILED DESCRIPTION:
The Internet has become an important tool for many people with health concerns [1,2] specially for adolescents [3,4]. Concerns about confidentiality, coupled with the stigma and shame associated with some conditions, specially sexually transmitted infections and other Health related problems make the internet a safe enviroment for adolescents to seek for information. This is thought to lead to an under-utilization of traditionally providers as the primary care health services.

These consultations, often made by young people, include sexual and reproductive health problems [5] and mental health disorders [6]. This can be a major problem, since the under-utilization of primary care services for certain topics and the search for advice on the Internet that is not usually trusted can subsequently lead to health complications that may require more expensive specialized medical interventions. long-term and, therefore, can translate into an increase in healthcare costs [7].

School programmes as Salut i Escola, have had as an objective all these years, to provide a more readily access to health care practitioners in order to improve their health related problems, doubts in sexual orientation, mental Health issues, drug related consultations and prevention of high-risk sexual behaviors by collaboration with educational centers and the community health services present in the territory.

Nowadays, with all the Advanced Technology we dispose, and because of the enormous amount of unstructured online content and the importance and difficulty of determining health information quality[8], it is almost obligatory to try to provide access to verified and make this study a tool to engage with adolescents and rovide them with accedd to trustful information.

Therefore, the Salut i Escola program together with the software of a well known company AGH Health, have been tried to minimize hesitation in seeking health advice through a chat application called Xatjove [9]. This is an asynchronous mobile text-based communication agent that connects users with healthcare professionals. These professionals provide appropriate guidance and advice to users in order to help them take Health related decisions.

As an anonymous digital health intervention, XatJove has the potential to address cost ineffectiveness caused by under-utilization health services in terms of shameful and stigmatized disorders.

According to a pilot study on e-Consultation (then known as WebGP), some of the top ten reasons for consultation of patients using this virtual tool included cystitis and problems with contraception (in women) [10]. It is known that if ignored, these conditions can lead to more serious, unwanted and costly complications (lack of contraception can lead to unwanted pregnancies and sexually transmitted infections) [11,12]. The fact that users routinely reported these problems through interventions health services such as e-Consultation is a positive sign in terms of an increased use of health services for sensitive but important conditions.

At the current time of the health crisis caused by the Covid-19 pandemic and to reduce the risk of infection, it makes more sense than ever to try to avoid face-to-face consultations of nursing professionals in institutes and also the visits of young people. to Primary Care Centers (CAPs). Great care must be taken that this does not mean a reduction in consultations on topics related to the health and school program. In addition, the health crisis is expected to lead to an increase in the need for emotional support by young people and agile tools are needed that use technologies that this sector of the population dominates and uses on a regular basis [13].

A sample of students aged 12 to 16 years from middle school and high school in the sanitary regions of the Anoia and Osona, province of Barcelona in the acadèmic course of 2020-2021.

A confidentiality form will be filled by every person partisipating in the study.

The parent or guardian of every student signed an informed consent document that described the purpose and procedure of the study. Students also signed separate assent forms with similar information.

Study design Quasi-experimental design were the data collected by our coustomised close-end survey, initial registration of the participants and the number of visits will be collected for further data analysis.

Place and Period of the Study Demografic region of Anoia and Osona, Barcelona. Duration of the study: Academic course of 2020-2021.

ELIGIBILITY:
Inclusion Criteria:

* All Anoia Students aged 12 to 16 years from middle school and high school

Exclusion Criteria:

* no

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-10-11 (Estimated)

PRIMARY OUTCOMES:
Survey | eigtht months
  Anoia students survey response of 6 multiple options and will be asked to rate on a scale of 1 to 10, the satisfaction of the service provided.

CONTACTS AND LOCATIONS:
Locations (1):
- SAP Anoia, Igualada, Barcelona, Spain

REFERENCES:
- [Derived] Sauch Valmana G, Vidal-Alaball J, Garcia Furio V, Testoni G, Espelt A, Exposito K, Saigi-Rubio F, Carre N, Sanz I, Vicens V. An Asynchronous, Mobile Text-Based Platform (XatJove Anoia) for Providing Health Services to Teenagers: Protocol for a Quasiexperimental Study. JMIR Res Protoc. 2021 Feb 3;10(2):e25062. doi: 10.2196/25062. PMID 33533729